CLINICAL TRIAL: NCT00420992
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Efficacy Study of Kadian NT (Morphine Sulfate Plus Naltrexone Hydrochloride Extended-Release) Capsules in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Hip or Knee
Brief Title: A Study of Embeda (Kadian NT, ALO-01) in Subjects With Pain Due to Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALO-KNT-301
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Results first posted 2009-10-30 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis; Chronic Pain
Keywords: hip; knee; pain; osteoarthritis; OA; Kadian; Alpharma; naltrexone; Opioid; morphine; Embeda; ALO-01
MeSH Terms: conditions — Osteoarthritis; Chronic Pain; Pain | interventions — morphine, naltrexone combination; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ALO-01 (Experimental): Up to 80 mg twice a day (bid)
  Interventions: Drug: ALO-01 (Morphine Sulfate Plus Naltrexone Hydrochloride Extended Release)
- Placebo (Placebo Comparator): Twice a day (bid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALO-01 (Morphine Sulfate Plus Naltrexone Hydrochloride Extended Release) — capsules, up to 80 mg bid
  Other Names: Embeda
  Arms: ALO-01
Drug: Placebo — capsules, bid
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Kadian NT (ALO-01) compared with placebo for treating moderate to severe chronic pain over a 12 week period.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of ALO-01 compared with placebo for the treatment of chronic moderate to severe pain (focusing on osteoarthritis of the hip or knee) as measured by mean change in diary Brief Pain Inventory (BPI) score of average pain (daily scores of average pain averaged over 7 days) from randomization to 12 weeks following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 21 years of age or older
* Subject is either not of childbearing potential OR subject must use an acceptable method of birth control if of childbearing potential
* Negative pregnancy test if female of childbearing potential
* Subject is in general good health
* Subject required treatment of joint pain within the last 90 days
* Subject has primary diagnosis of osteoarthritis (OA) of the hip or knee

Exclusion Criteria:

* Subject has a documented history of allergic reaction or intolerance to morphine or other opioids
* Subject is pregnant or breast-feeding
* Subject is receiving systemic chemotherapy
* Subject has a history of drug abuse/dependence/misuse or alcohol abuse/dependence
* Subject has history of major depressive disorder not controlled with medication
* Subject has any chronic pain syndrome (i.e., fibromyalgia) that may interfere with the symptoms of OA
* Subject has active gastrointestinal disease, with the exception of gastroesophageal reflux disease (GERD)
* Subject has a documented history of rheumatoid arthritis, uncontrolled inflammatory arthritis or non-steroidal anti-inflammatory drug (NSAID)-dependent inflammatory arthritis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B. Jones, MD, PharmD, Study Director — Alpharma Pharmceuticals
Locations (80):
- United States (80):
  - The Birmingham Pain Center, Birmingham, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Arizona Center for Clinical Research, Peoria, Arizona
  - Arizona Research Center, Inc, Phoenix, Arizona
  - Premiere Pharmaceutical Research, LLC, Tempe, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Anaheim, California
  - STAT-CARE / Crest Clinical Trials, Anaheim, California
  - Southbay Pharma Research, Buena Park, California
  - Providence Clinical Res. (C-trials), Burbank, California
  - Med Investigators Inc, Fair Oaks, California
  - Quality of Life Medical Center, LLC, Hawaiian Gardens, California
  - NervePro Research, Irvine, California
  - UCSD Pain and Palliative Care, La Jolla, California
  - USCD Pain and Palliative Care, La Jolla, California
  - Private Practice, Pico Rivera, California
  - Pain Institute of Santa Monica, Santa Monica, California
  - Boling Clinical Trials, Upland, California
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - MD Clinical, Hallandale, Florida
  - Eastern Research, Hialeah, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institiute, Jupiter, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Innovative Research of West Florida, Largo, Florida
  - Pharmaceutical Research Associates Inc, Merritt Island, Florida
  - Ormond Medical Arts - Pharmaceutical Research Center, Ormond Beach, Florida
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Gold Coast Research LLC, Weston, Florida
  - River Birch Research Alliance, Blue Ridge, Georgia
  - Best Clinical Research, Decatur, Georgia
  - Non-Surgical Orthopaedic and Spine Center, Marietta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Research Associates of Central Illinois, Peoria, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Welborn Clinic, Newburgh, Indiana
  - International Clinical Research Institute, Inc, Overland Park, Kansas
  - Clinical Trials Management, LLC, Mandeville, Louisiana
  - Lousiana Research Associates Inc., New Orleans, Louisiana
  - Internal Research Center, Towson, Maryland
  - Phase III Clinical Research, Fall River, Massachusetts
  - Northeast Medical Research Associates, Inc, No Dartmouth, Massachusetts
  - FutureCare Studies, Springfield, Massachusetts
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - Medex Healthcare Research Inc, St Louis, Missouri
  - Lovelace Scientific, Henderson, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Partners in Primary Care, Voorhees Township, New Jersey
  - Elkind Headache Center, Mount Vernon, New York
  - The Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Clinical Research Source, Inc, Toledo, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - LVH Neurosciences and Pain Research, Allentown, Pennsylvania
  - Pennsylvania Research Institute, Bensalem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Commonwealth Primary Care / Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Pivotal Clinical Research, LLC, Souderton, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - Premier Medical Group, Clarksville, Tennessee
  - SCRI, Cordova, Tennessee
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - SCRI, Memphis, Tennessee
  - Integrity Clinical Research, LLC, Milan, Tennessee
  - Walter F. Chase, MD, PA, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Team Research of Central Texas, Killeen, Texas
  - Radiant Research, San Antonio Northeast, San Antonio, Texas
  - North San Antonio Healthcare Associates, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - HypotheTest, LLC, Roanoke, Virginia

REFERENCES:
- [Derived] Setnik B, Pixton GC, Webster LR. Safety profile of extended-release morphine sulfate with sequestered naltrexone hydrochloride in older patients: pooled analysis of three clinical trials. Curr Med Res Opin. 2016;32(3):563-72. doi: 10.1185/03007995.2015.1131153. Epub 2016 Jan 26. PMID 26695349

RESULTS

PARTICIPANT FLOW:
Period: Titration Phase
Arm/Group | ALO-01 | Placebo
Started | 547 (All patients received ALO-01 during open-label titration phase) | 0
Completed | 344 | 0
Not Completed | 203 | 0
Period: Maintenance Phase
Arm/Group | ALO-01 | Placebo
Started | 171 | 173
Completed | 110 | 98
Not Completed | 61 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALO-01 | Placebo | Total
Number analyzed (Participants) | 171 | 173 | 344
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.62) | 54.7 (12.92) | 54.4 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 95 | 201
  Male | 65 | 78 | 143

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomization to 12 Weeks Following Randomization in Diary Brief Pain Inventory Score of Average Pain (Daily Scores of Average Pain Averaged Over 7 Days)
Description: Change in pain intensity scale. Average pain intensity over last 24 hours rated daily from 0=no pain to 10=worst pain.
Time Frame: randomization to 12 weeks following randomization
Population: intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | ALO-01 | Placebo
Number analyzed (Participants) | 170 | 173
units on scale | -0.2 (1.94) | 0.3 (2.05)
Statistical Analysis 1: Comparison: ALO-01 vs Placebo; Null hypothesis: mean change from baseline is the same for ALO-01 and placebo; Test type: Superiority or Other; p = 0.0445, ANCOVA — Threshold for statistical significance: P=0.05. No adjustment for multiple comparisons necessary; Model included treatment as factor and baseline pain score as covariate

ADVERSE EVENTS:
Groups:
- Titration ALO-01: Open-label ALO-01
Arm/Group | ALO-01 | Placebo | Titration ALO-01
Serious Adverse Events (participants affected / at risk) | 6/171 | 3/173 | 3/547
Other Adverse Events (participants affected / at risk) | 54/171 | 48/173 | 301/547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALO-01 (N=171) | Placebo (N=173) | Titration ALO-01 (N=547)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALO-01 (N=171) | Placebo (N=173) | Titration ALO-01 (N=547)
Constipation (Gastrointestinal disorders) | 12 | 7 | 167
Diarrhoea (Gastrointestinal disorders) | 21 | 21 | 15
Nausea (Gastrointestinal disorders) | 20 | 13 | 115
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 31
Vomiting (Gastrointestinal disorders) | 12 | 4 | 50
Somnolence (Nervous system disorders) | 2 | 5 | 78
Dizziness (Nervous system disorders) | 3 | 3 | 47
Headache (Nervous system disorders) | 12 | 6 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 38
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the Sponsor for review. Sponsor may request a delay in publication to allow the filing of patent applications before publication or release. The sponsor can require deletion of Confidential Information or request correction of inaccuracies.